CLINICAL TRIAL: NCT01946061
Title: A Phase II Trial of Adjuvant Chemotherapy With S-1 Plus Oxaliplatin for Locally Advanced Gastric Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was stopped because of difficulties of supplying the drug.
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2013-0452
Record Dates: First submitted 2013-09-12; First posted 2013-09-19 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Advanced Gastric Cancer
Keywords: Oxaliplatin, S-1, Gastric cancer, Adjuvant chemotherapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — S 1 (combination); Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment group (Experimental)
  Interventions: Drug: S-1 plus oxaliplatin

INTERVENTIONS:
Drug: S-1 plus oxaliplatin — Patients will receive adjuvant chemotherapy of eight 3-week cycles of oral S-1 (70 mg/m2/day on days 1 to 14 of each cycle) plus intravenous oxaliplatin (130 mg/m2 on day 1 of each cycle) for 6 months after D2 gastrectomy.

SUMMARY:
Patients with advanced gastric cancer have showed poor prognosis. Only 81% of the patients could underwent curative surgery. In those, about 60% of patients would survive after 5 years from the surgery. As a result, role of chemotherapy has been increased. In ACTS-GC trial, S-1 adjuvant therapy after D2 gastrectomy increased overall survival rate in advanced gastric cancer patients. However, subgroup analysis showed that S-1 adjuvant therapy was insufficient in patients with stage III or IV (according to the AJCC 6th criteria) gastric cancer. In addition, CLASSIC trial demonstrated that oxaliplatin plus capecitabine adjuvant therapy could increase disease-free survival after D2 gastrectomy in advanced gastric cancer patients. Notwithstanding these trial, optimal adjuvant regimen of advanced gastric cancer has not been established. We aimed to evaluate efficacy of S-1 plus oxaliplatin as adjuvant chemotherapy after D2 gastrectomy in stage III (according to the AJCC 7th criteria) gastric cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Age, between 19 and 75
* Histologically proven advanced gastric cancer
* R0 resection after D2 gastrectomy
* Stage III (according to the AJCC 7th criteria)
* ECOG status 0 to 2

Exclusion Criteria:

* Malignancy history other than gastric cancer
* Previous chemotherapy history for gastric cancer
* Previous radiotherapy history for gastric cancer
* Pregnancy or breast milk feeding
* Grade 3 or more of neuropathy
* Active infection
* Severe hepatic dysfunction
* Severe renal dysfunction
* Severe bone marrow dysfunction
* Significant neurologic or psychologic disease
* Inadequate condition for receiving chemotherapy due to significant systemic disease
* Patients who receives drugs which can be interacted with S-1

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-05; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
3-year disease-free survival | 3 years from the surgery
  3-year disease-free survival will be assessed by imaging study including CT and PET.

CONTACTS AND LOCATIONS:
Locations (1):
- Severnace Hospital, Seoul, South Korea

REFERENCES:
- [Background] Sakuramoto S, Sasako M, Yamaguchi T, Kinoshita T, Fujii M, Nashimoto A, Furukawa H, Nakajima T, Ohashi Y, Imamura H, Higashino M, Yamamura Y, Kurita A, Arai K; ACTS-GC Group. Adjuvant chemotherapy for gastric cancer with S-1, an oral fluoropyrimidine. N Engl J Med. 2007 Nov 1;357(18):1810-20. doi: 10.1056/NEJMoa072252. PMID 17978289